CLINICAL TRIAL: NCT03063164
Title: A Prospective, Randomized, Fellow Eye Comparison of Fellow Eyes Undergoing LASIK With the Intralase IFS150 Versus the Visumax
Brief Title: A Comparison of LASIK Outcomes Using Two Femtosecond Lasers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward E. Manche (Other)
Responsible Party: Sponsor-Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33356
Record Dates: First submitted 2017-02-11; First posted 2017-02-24 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Myopia; Astigmatism
Keywords: Femtosecond laser; Visumax; Intralase IFS150; LASIK
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Eye to eye comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intralase IFS (Active Comparator): Intralase IFS vs. Visumax
  Interventions: Device: Intralase IFS150
- Visumax (Active Comparator): Visumax vs. Intralase iFS
  Interventions: Device: Visumax

INTERVENTIONS:
Device: Intralase IFS150 — Intralase flap creation
  Arms: Intralase IFS
Device: Visumax — Visumax flap creation
  Arms: Visumax

SUMMARY:
Comparing LASIK outcomes using two femtosecond lasers

DETAILED DESCRIPTION:
Patients will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the patient from the study, then the investigator will inform the patient and make an appropriate referral. Patients deemed appropriate for the study after a comprehensive examination including computerized videokeratography can be enrolled. Patients will undergo bilateral simultaneous eye surgery. Which eye is treated with the Intralase IFS 150 and which eye is treated with VisuMax will be randomized so there is a 50% chance for either eye to receive one treatment. Patients will be seen on the day of surgery, post op day one, one month, three months, six months and one year. Patients will receive topical antibiotics in each eye for one week following the procedure. Patients will receive pred forte 1% ophthalmic drops for one week after treatment. Patients will also receive vigamox ophthalmic drops for four days after treatment. All of this is within the usual and customary standard of care for the treatment of patients undergoing LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes. Nearsightedness between -0.25 diopters and -11.00 diopters with or without astigmatism of up to 5.00 diopters.

Exclusion Criteria:

* Subjects under the age of 21
* Subjects over the age of 60
* Subjects with corneal ectatic disorders

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Intralase IFS Eye; Visumax Eye: Participants received treatment with Intralase IFS in one eye and treatment with Visumax in their fellow eye.
Period: Overall Study
Arm/Group | Intralase IFS Eye | Visumax Eye
Started | 7; 7 Eyes | 7; 7 Eyes
Completed | 7; 7 Eyes | 7; 7 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- All Participants: Participants received treatment with Intralase IFS in one eye and treatment with Visumax in their fellow eye.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Number analyzed (Eyes) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Caucasian | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: ETDRS Uncorrected Visual Acuity
Description: Number of eyes with an uncorrected visual acuity of 20/20 at 12 months measured using ETDRS testing charts
Time Frame: At post-operative month 12
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 7 | 7
Number analyzed (Eyes) | 7 | 7
Eyes | 5 | 5

2. Secondary Outcome: Anterior Segment Ocular Coherence Tomography Measurement of Flap Thickness
Description: Anterior segment ocular coherence tomography
Time Frame: At postoperative month one
Population: Data were corrupted and could not be analyzed
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cochet Bonnet Asthesiometry Measurement of Corneal Sensation
Description: Cochet Bonnet Asthesiometry is measured on a scale of 1-6. Scores of 5 and above are considered normal.
Time Frame: At postoperative month twelve
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 7 | 7
Number analyzed (Eyes) | 7 | 7
Eyes
  Score of greater than or equal to 5 | 7 | 7
  Score of less than 5 | 0 | 0

4. Secondary Outcome: Best Spectacle Corrected Visual Acuity
Description: Number of eyes losing 2 or more lines of corrected distance visual acuity measured by ETDRS testing charts
Time Frame: Postoperative month 12
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 7 | 7
Number analyzed (Eyes) | 7 | 7
Eyes | 0 | 0

5. Secondary Outcome: Aberrometry
Description: Aberrometry images will be obtained on the iDesign aberrometer
Time Frame: One three, six and twelve months
Population: The data were corrupted and could not be analyzed
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Questionnaire Measuring Patient Preference for Laser Device
Description: Participants were asked if they preferred having LASIK surgery with either the Visumax laser, the Intralase iFS laser or had no preference between the two lasers.
Time Frame: Intraoperative (Approximately 1 minute after completion of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 7
Participants
  Preferred Visumax | 3
  Preferred Intralase IFS | 2
  No preference | 2

7. Secondary Outcome: Patient Reported Outcomes With LASIK
Description: PROWL study questionnaire
Time Frame: One month, three months, six months and twelve months
Population: Questionnaire data were corrupted and could not be analyzed.
Arm/Group | Intralase IFS Eye | Visumax Eye
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Twelve months
Description: Data on all serious and non-serious Adverse Events experienced by participants were collected, irrespective of the event's relation to the treated eye.
Arm/Group | Intralase IFS Eye | Visumax Eye
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
The study did not meet its planned enrollment number

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03063164/Prot_000.pdf